CLINICAL TRIAL: NCT07053189
Title: Effects of Interproximal Reduction and Attachment Application on Effectiveness of Rotational Tooth Movement in Clear Aligner Therapy
Brief Title: Evaluation of IPR and Attachments on Rotational Tooth Movement in Clear Aligner Therapy
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Aylin Alaçam, Asis.Prof.,Lokman Hekim University, Faculty of Dentistry, Department of Orthodontics, Lokman Hekim University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB No: 100/050/REK.001
Record Dates: First submitted 2025-05-21; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Malocclusion; Displaced or Missing Teeth
Keywords: rotation; interproximal enamel reduction; attachment; clear aligner therapy; effectiveness
MeSH Terms: conditions — Malocclusion; Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Rotational tooth movement in clear aligner therapy (Experimental)
  Interventions: Device: Clear Aligner treatment

INTERVENTIONS:
Device: Clear Aligner treatment — Interproximal enamel reduction and attachment impact

SUMMARY:
This study is testing whether clear aligners (Invisalign®) can help fix teeth that are rotated. The researchers want to learn if using two common methods-interproximal enamel reduction (IPR) and attachments-makes rotation correction more successful.

Participants in the study will wear custom-made aligners for about 20 to 22 hours every day. They will switch to a new set of aligners every 2 weeks.

The study will look at tooth movement over time by using a digital planning tool called ClinCheck®, which helps plan and measure how much teeth have moved.

The researchers want to answer three main questions:

Do Invisalign® aligners work well for correcting rotated teeth?

Does IPR help improve rotation correction?

Do attachments help improve rotation correction?

The goal is to understand whether these tools work better together or separately to move teeth into better alignment.

DETAILED DESCRIPTION:
This study is about clear aligners, which are plastic trays that gently move teeth. The researchers want to know how well aligners can fix teeth that are rotated (turned out of their normal position). They also want to test whether two common tools-interproximal enamel reduction (IPR) and attachments-help aligners work better when correcting rotated teeth.

IPR means gently shaving a small amount of enamel between teeth to make space for movement.

Attachments are small, tooth-colored bumps added to teeth to help the aligners grip better and apply more force.

The study includes 35 participants who are being treated with Invisalign® clear aligners. All of them have full adult teeth (except wisdom teeth), mild to moderate crowding, and a type of bite called Class I malocclusion.

Participants wear their aligners for 20 to 22 hours a day, changing to a new set every 2 weeks. The average treatment includes about 18 aligners.

Each participant had a digital scan of their teeth taken at the beginning using an iTero Element® scanner. This scan was used to design a personalized treatment plan using ClinCheck® software, which predicts how the teeth should move.

During treatment, researchers place:

Rectangular attachments on some front and back teeth to improve control

Optimized attachments on teeth that are rotated more than 0.5°, especially premolars and canines

ELIGIBILITY:
Inclusion Criteria:

Adults with full permanent dentition (excluding wisdom teeth)

Angle Class I malocclusion

Mild to moderate crowding in the upper and lower arches

Planned treatment with clear aligners for both jaws

Rotated teeth within the correction limits recommended by Align Technology®

Willing and able to wear aligners for 20-22 hours per day

Able to attend follow-up visits every 2 aligners (~4 weeks)

-

Exclusion Criteria:

Previous orthodontic treatment

Need for additional orthodontic appliances (e.g., elastics or rubber bands)

Periodontal disease or other active oral health problems

Presence of prosthetic dental work (e.g., crowns or bridges)

Need for tooth extraction during aligner treatment

Medical conditions that may interfere with orthodontic treatment compliance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in tooth rotation (degrees) from baseline (T0) to refinement (T1), measured from Clincheck software | 36,9 weeks
  Comparison of tooth rotation correction with IPR and attachments

CONTACTS AND LOCATIONS:
Locations (1):
- A special dental clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Protect personal data